CLINICAL TRIAL: NCT07202832
Title: Efficacy and Safety of Urine Alkalinization in Treatment of Uncomplicated Urinary Tract Infection in Women: A Randomized Controlled Trial
Brief Title: Urine Alkalinization for UTI in Women: RCT
Acronym: UTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Esam Saad Mohamed Darwish, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PreIRB-Assiut-URO002
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: UTI - Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Potassium Citrate; Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Citrate Treatment for UTI Symptom Relief (Active Comparator): Participants in this arm will receive potassium citrate oral sachets twice daily for 7 days. The aim is to assess the effectiveness of potassium citrate in alleviating UTI symptoms such as dysuria and urgency in women with uncomplicated urinary tract infections. Participants will be monitored for symptom improvement, side effects, and any changes in urine culture.
  Interventions: Drug: potassium citrate
- Nitrofurantoin Antibiotic Treatment for UTI (Active Comparator): Participants in this group will receive the antibiotic "Nitrofurantoin" for 7 days. This group serves as a control to compare the effectiveness of antibiotics against urinary alkalinization in treating symptoms of uncomplicated urinary tract infections (UTIs). The primary outcomes include symptom relief, changes in urine culture, and the occurrence of any side effects. This group's results will be compared with Arm 1 to determine if urinary alkalinization is equally or more effective than antibiotics in managing UTI symptoms.
  Interventions: Drug: Nitrofurantoin

INTERVENTIONS:
Drug: potassium citrate — Potassium citrate is a medication used to alkalinize the urine, providing symptomatic relief of dysuria in patients with urinary tract infections (UTIs). In this study, participants in Arm 1 will receive potassium citrate for a period of 7 days. The treatment is aimed at reducing discomfort related to UTIs, such as burning sensations during urination and suprapubic pain. In addition to symptomatic relief, the intervention may also enhance bacterial phagocytosis and bacterial killing in the urine. Participants will be monitored for any side effects or adverse events during the treatment period.
  Arms: Potassium Citrate Treatment for UTI Symptom Relief
Drug: Nitrofurantoin — Nitrofurantoin is an antibiotic commonly used to treat uncomplicated urinary tract infections (UTIs). In this arm, participants will receive Nitrofurantoin for 7 days to treat their UTI. The primary objective is to evaluate its effectiveness in reducing UTI symptoms, such as dysuria, urgency, frequency, and suprapubic discomfort. This intervention will be compared with the urinary alkalinization therapy used in Arm 1. Researchers will also monitor changes in urine culture and any adverse events related to the antibiotic treatment.
  Arms: Nitrofurantoin Antibiotic Treatment for UTI

SUMMARY:
The goal of this clinical trial is to evaluate whether urinary alkalinization using potassium citrate can relieve symptoms and improve urine culture results in women aged 18 to 50 years with uncomplicated urinary tract infections (UTIs). The main questions it aims to answer are:

Does urinary alkalinization reduce UTI symptom scores by Day 7?

Does it lead to better urine culture results compared to antibiotic?

Researchers will compare urinary alkalinization with potassium citrate to antibiotic to see if it provides more symptom relief and better microbiological outcomes.

Participants will:

Take either potassium citrate or antibiotic

Be assessed for symptoms and adverse events on Day 7

Provide a urine sample for culture before and after treatment

Report any return visits due to worsening symptoms or medication side effects

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 and ≤ 50.
* Symptoms of uncomplicated UTI or cystitis; including urinary frequency, urgency and dysuria.
* Positive urine culture of mid-urine urine.

Exclusion Criteria:

* Post menopausal women.
* Pregnancy.
* Complicated UTIs, such as those requiring hospital admission, infections associated with fevers, those with urinary tract abnormalities, urinary tract calculi or urinary tract obstruction.
* History of recurrent UTI.
* Recent antibiotic use.
* Acute pyelonephritis.
* Immunocompromising conditions.
* Chronic conditions such as interstitial cystitis, painful bladder syndrome, chronic pelvic pain syndrome.
* Patients with CKD.
* Patients with allergy to potassium citrate.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Relief (Dysuria, Urgency, and Frequency) in UTI Patients Treated with Potassium Citrate vs. Nitrofurantoin | 7 days (Participants will be assessed at baseline, day 3, and day 7).
  The primary outcome of this study is the reduction in urinary tract infection (UTI) symptoms, specifically dysuria (painful urination), urgency, and frequency, after 7 days of treatment with either Potassium Citrate or Nitrofurantoin. The severity of these symptoms will be measured using a standardized symptom questionnaire, where participants will rate the intensity of their symptoms at baseline (pre-treatment), day 3, and day 7. A reduction of ≥50% in symptom severity will be considered clinically significant. The results will be compared between the Potassium Citrate and Nitrofurantoin groups to determine which treatment is more effective in relieving UTI symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Darwish, Lecturer, Principal Investigator — Urology Department, Faculty of Medicine, Assiut University
Locations (1):
- Urology Department, Faculty of Medicine, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No